CLINICAL TRIAL: NCT05776108
Title: A Phase 1, Single-center, Randomized, Open-label, Single Dose, Three-period, Balanced Crossover Study to Assess the Effect of Food on the Pediatric Dispersible Tablet Formulation of Cabotegravir and to Assess the Relative Bioavailability Between the Pediatric Dispersible Tablet (DT) Formulation and Immediate Release (IR) Tablet Formulation of Cabotegravir in Healthy Adult Participants
Brief Title: A Study to Assess the Food Effect and the Relative Bioavailability of the Cabotegravir (CAB) Pediatric Dispersible Tablet (DT) Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 219679
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: HIV Infections
Keywords: Bioavailability; Cabotegravir; Dispersible tablet; Food effect; Human immunodeficiency virus; Immediate release tablet
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Masking Description: This is an open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CAB IR Formulation (reference)/CAB DT Formulation (Test 1)/CAB DT Formulation (Test 2) (Experimental): Participants will receive CAB IR Formulation (reference) under fasted conditions in treatment period 1 followed by CAB DT Formulation (test 1) under fasted conditions in treatment period 2 followed by CAB DT Formulation (test 2) under fed conditions in treatment period 3. There will be a minimum washout period of 14 days between each treatment .
  Interventions: Drug: Cabotegravir IR Formulation (reference); Drug: Cabotegravir DT Formulation (test 1); Drug: Cabotegravir DT Formulation (test 2)
- CAB DT Formulation (Test 1)/CAB IR Formulation (reference)/CAB DT Formulation (test 2) (Experimental): Participants will receive CAB DT Formulation (test 1) under fasted conditions in treatment period 1 followed by CAB IR Formulation (reference) under fasted conditions in treatment period 2 followed by CAB DT Formulation (test 2) under fed conditions in treatment period 3. There will be a minimum washout period of 14 days between each treatment.
  Interventions: Drug: Cabotegravir IR Formulation (reference); Drug: Cabotegravir DT Formulation (test 1); Drug: Cabotegravir DT Formulation (test 2)
- CAB DT Formulation (test 2)/CAB IR Formulation (reference)/CAB DT Formulation (test 1) (Experimental): Participants will receive CAB DT Formulation (test 2) under fed conditions in treatment period 1 followed by CAB IR Formulation (reference) under fasted conditions in treatment period 2 followed by CAB DT Formulation (test 1) under fasted conditions in treatment period 3. There will be a minimum washout period of 14 days between each treatment.
  Interventions: Drug: Cabotegravir IR Formulation (reference); Drug: Cabotegravir DT Formulation (test 1); Drug: Cabotegravir DT Formulation (test 2)
- CAB IR Formulation (reference)/CAB DT Formulation (test 2)/CAB DT Formulation (test 1) (Experimental): Participants will receive CAB IR Formulation (reference) under fasted conditions in treatment period 1 followed by CAB DT Formulation (test 2) under fed conditions in treatment period 2 followed by CAB DT Formulation (test 1) under fasted conditions in treatment period 3. There will be a minimum washout period of 14 days between each treatment.
  Interventions: Drug: Cabotegravir IR Formulation (reference); Drug: Cabotegravir DT Formulation (test 1); Drug: Cabotegravir DT Formulation (test 2)
- CAB DT Formulation (test 1)/CAB DT Formulation (test 2)/CAB IR Formulation (reference) (Experimental): Participants will receive CAB DT Formulation (test 1) under fasted conditions in treatment period 1 followed by CAB DT Formulation (test 2) under fed conditions in treatment period 2 followed by CAB IR Formulation (reference) under fasted conditions in treatment period 3. There will be a minimum washout period of 14 days between each treatment.
  Interventions: Drug: Cabotegravir IR Formulation (reference); Drug: Cabotegravir DT Formulation (test 1); Drug: Cabotegravir DT Formulation (test 2)
- CAB DT Formulation (test 2)/CAB DT Formulation (test 1)/CAB IR Formulation (reference) (Experimental): Participants will receive CAB DT Formulation (test 2) under fed conditions in treatment period 1 followed by CAB DT Formulation (test 1) under fasted conditions in treatment period 2 followed by CAB IR Formulation (reference) under fasted conditions in treatment period 3. There will be a minimum washout period of 14 days between each treatment.
  Interventions: Drug: Cabotegravir IR Formulation (reference); Drug: Cabotegravir DT Formulation (test 1); Drug: Cabotegravir DT Formulation (test 2)

INTERVENTIONS:
Drug: Cabotegravir IR Formulation (reference) — Cabotegravir IR Formulation (reference) will be administered.
Drug: Cabotegravir DT Formulation (test 1) — Cabotegravir DT Formulation (test 1) will be administered.
Drug: Cabotegravir DT Formulation (test 2) — Cabotegravir DT Formulation (test 2) will be administered.

SUMMARY:
This study will assess the relative bioavailability of the CAB DT formulation relative to that of the CAB IR formulation and to assess the effect of food on the CAB DT formulation.

ELIGIBILITY:
Inclusion criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent form (ICF).
* Participants who are healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring (history and electrocardiogram).
* Body weight greater than or equal to (>=) 50.0 kilograms (kg) (110 pounds [lbs]) for males and >= 45 kg (99 lbs) for females and Body mass index within the range 18.5 to 31.0 kilogram per meter square (kg/m2) (inclusive) at Screening.
* Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  * Female: A female participant is eligible to participate if she is not pregnant or breastfeeding and is a Women of non child bearing potential (WONCBP) OR Is a Women of child bearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of less than (<)1 percent (%) per year).
  * A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention (i.e., Day-1 of each treatment Period)
  * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* History of seizures, and participants are required to have been seizure free, off anti epileptic drugs for a minimum of 2 years and will only be considered for enrollment following discussion with the Medical Monitor
* Abnormal blood pressure as determined by the investigator.
* Medical history of cardiac arrhythmias, prior myocardial infarction in the past 3 months, or cardiac disease or a family or personal history of long QT syndrome.
* A pre-existing condition interfering with normal gastrointestinal anatomy or motility (e.g., gastroesophageal reflux disease, gastric ulcers, gastritis), hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study intervention.
* Known suspected active Coronavirus disease 2019 (COVID-19) infection OR contact with an individual with known COVID-19 , within 14 days of study enrollment
* Any acute laboratory abnormality at screening which, in the opinion of the investigator, should preclude participation in the study of an investigational compound.
* Any Grade 2 to 4 laboratory abnormality at screening, with Creatine Phosphokinase and lipid abnormalities (e.g., total cholesterol, triglycerides), and ALT abnormalities, will exclude a participant from the study unless the investigator can provide a compelling explanation for the laboratory result(s) and has the assent of the sponsor.
* A positive test result for drugs of abuse (including marijuana), alcohol, or tobacco (indicating active current smoking) at screening or before the first dose of study intervention.
* Unable to refrain from the use of prescription or non-prescription drugs as detailed in the protocol.
* Unwillingness to abstain from excessive consumption of any food or drink detailed in the protocol.
* Would not be able to accommodate the blood loss during participation in the study
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* Current enrollment or past participation in another investigational study as detailed in the protocol.
* Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing. - Current enrollment or past participation in this clinical study.
* Positive hepatitis B and/or C test result at screening or within 3 months prior to first dose of study intervention.
* Positive pre-study drug/alcohol screen, including Tetrahydrocannabinol
* Positive Human immunodeficiency virus (HIV) antibody test (4th generation assay required).
* Regular use of tobacco- or nicotine-containing products within 6 months prior to screening
* History of regular alcohol consumption within 6 months of the study,
* History of sensitivity, prior intolerance or hypersensitivity to any of the study interventions, or components thereof, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Participant and/or his her family is part of sponsor, clinical site, third party personnel.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-inf]) following administration of CAB DT after a high fat meal | Up to 168 hours
Area under the concentration time curve from time zero (pre-dose) extrapolated to last time of quantifiable concentration (AUC[0-last]) following administration of CAB DT after a high fat meal | Up to 168 hours
Maximum observed concentration (Cmax) following administration of CAB DT after a high fat meal | Up to 168 hours
AUC(0-inf) following administration of CAB DT in fasted state | Up to 168 hours
AUC(0-last) following administration of CAB DT in fasted state | Up to 168 hours
Cmax following administration of CAB DT in fasted state | Up to 168 hours
AUC(0-inf) following administration of CAB IR in fasted state | Up to 168 hours
AUC(0-last) following administration of CAB IR in fasted state | Up to 168 hours
Cmax following administration of CAB IR in fasted state | Up to 168 hours

SECONDARY OUTCOMES:
Apparent terminal phase half-life (T1/2) following administration of CAB DT | Up to 168 hours
Lag time before observation of drug concentrations in sampled matrix (tlag) following administration of CAB DT | Up to 168 hours
Time of occurrence of Cmax (Tmax) following administration of CAB DT | Up to 168 hours
Area under the concentration time curve from time zero extrapolated to 72 hours post-dose AUC(0-72) following administration of CAB DT | Up to 72 Hours
Concentration at 24 hours post-dose (C24) of following administration of CAB DT | At 24 Hours
Apparent oral clearance (CL/F) following administration of CAB DT | Up to 168 hours
Apparent volume of distribution (Vz/F) following administration of CAB DT | Up to 168 hours
T1/2 following administration of CAB DT in fasted state | Up to 168 hours
Tlag following administration of CAB DT in fasted state | Up to 168 hours
Tmax following administration of CAB DT in fasted state | Up to 168 hours
AUC(0-72) following administration of CAB DT in fasted state | Up to 72 Hours
C24 following administration of CAB DT in fasted state | At 24 Hours
CL/F following administration of CAB DT in fasted state | Up to 168 hours
Vz/F following administration of CAB DT in fasted state | Up to 168 hours
T1/2 following administration of CAB IR in fasted state | Up to 168 hours
Tlag following administration of CAB IR in fasted state | Up to 168 hours
Tmax following administration of CAB IR in fasted state | Up to 168 hours
AUC(0-72) following administration of CAB IR in fasted state | Up to 72 Hours
C24 following administration of CAB IR in fasted state | Up to 168 hours
CL/F following administration of CAB IR in fasted state | Up to 168 hours
Vz/F following administration of CAB IR in fasted state | Up to 168 hours
Number of participants with Non-Serious Adverse events (AEs) and Serious adverse events (SAEs) | Up to 6 Weeks
Number of participants with AEs by severity | Up to 6 Weeks
Change from Baseline in Vital sign parameter: Oral Temperature (Degrees Celsius) | Baseline and Up to 6 Weeks
Change from Baseline in Vital sign parameter: Pulse rate (Beats per minute) | Baseline and Up to 6 Weeks
Change from Baseline in Vital sign parameter: Respiratory rate (Breaths per minute) | Baseline and Up to 6 Weeks
Change from Baseline in Vital sign parameter: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) (Millimeters of mercury) | Baseline and Up to 6 Weeks
Change from Baseline in Electrocardiogram (ECG) parameters: PR Interval, QRS Interval, QT Interval, Corrected QT interval using the Fridericia formula (QTcF) (Milliseconds) | Baseline and Up to 6 Weeks
Number of participants with maximum toxicity grade increase from Baseline in hematology, chemistry and urinalysis parameters | Baseline and Up to 6 Weeks
Change from Baseline in hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet Count (Giga cells per Liter) | Baseline and Up to 6 Weeks
Change from Baseline in hematology parameter: Red Blood Cell Count (Trillion cells per liter) | Baseline and Up to 6 Weeks
Change from Baseline in hematology parameter: Hemoglobin (Grams per liter) | Baseline and Up to 6 Weeks
Change from Baseline in hematology parameter: Hematocrit (Proportion of red blood cells in blood) | Baseline and Up to 6 Weeks
Change from Baseline in hematology parameter: Mean Corpuscular Volume (Femtoliters) | Baseline and Up to 6 Weeks
Change from Baseline in hematology parameter: Mean Corpuscular Hemoglobin (Picograms) | Baseline and Up to 6 Weeks
Change from Baseline in hematology parameter: Percentage of Reticulocytes (Percentage of reticulocytes) | Baseline and Up to 6 Weeks
Change from Baseline in chemistry parameters: Creatinine, Total and Direct Bilirubin (Micromoles per liter) | Baseline and Up to 6 Weeks
Change from Baseline in chemistry parameters: Calcium, Glucose, Potassium, Sodium, Blood urea nitrogen, Carbon dioxide (Millimoles per liter) | Baseline and Up to 6 Weeks
Change from Baseline in chemistry parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP), Aspartate Aminotransferase (AST), and Creatine phosphokinase (International units per liter) | Baseline and Up to 6 Weeks
Change from Baseline in chemistry parameters: Total Protein (Grams per liter) | Baseline and Up to 6 Weeks
Number of participants with abnormal urinalysis parameters | Up to 6 Weeks
Absolute values of hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils and Platelet Count (Giga cells per Liter) | Up to 6 Weeks
Absolute values of hematology parameter: Red Blood Cell Count (Trillion cells per liter) | Up to 6 Weeks
Absolute values of hematology parameter: Hemoglobin (Grams per liter) | Up to 6 Weeks
Absolute values of hematology parameter: Hematocrit (Proportion of red blood cells in blood | Up to 6 Weeks
Absolute values of hematology parameter: Mean Corpuscular Volume (Femtoliters) | Up to 6 Weeks
Absolute values of hematology parameter: Mean Corpuscular Hemoglobin (Picograms) | Up to 6 Weeks
Absolute values of hematology parameter: Percentage of Reticulocytes (Percentage of reticulocytes) | Up to 6 Weeks
Absolute values of chemistry parameters: Creatinine, Total and Direct Bilirubin (Micromoles per liter) | Up to 6 Weeks
Absolute values of chemistry parameters: Calcium, Glucose, Potassium, Sodium, Blood urea nitrogen, Carbon dioxide (Millimoles per liter) | Up to 6 Weeks
Absolute values of chemistry parameters: ALT, ALP, AST and Creatine phosphokinase (International units per liter) | Up to 6 Weeks
Absolute values of chemistry parameters: Total Protein (Grams per liter) | Up to 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/